CLINICAL TRIAL: NCT02040961
Title: Assessment of the the ETView Double-lumen Tube
Acronym: ETView1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: An incident, burned tube, happened before intubation. The promoter decided to stop the study.
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012/64; 2012-A01552-41 (Other: ANSM)
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Tracheal Intubation
Keywords: Patients; Undergoing; Elective; Thoracic; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EtView (Experimental): Use of ETVew double-lumen tube
  Interventions: Device: ETView Double-Lumen Tube

INTERVENTIONS:
Device: ETView Double-Lumen Tube — Tracheal intubation is performed using a ETView Double-Lumen Tube

SUMMARY:
The double tube ETView is particularly innovative as it includes an integrated optical fiber to visualize the carena. This study aims to verify if if its use avoids the requirement of a fibreoptic bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* elective thoracic surgery with anticipated use of a DLT

Exclusion Criteria:

* left pneumonectomy or left lobectomy requiring an anastomosis on the left main bronchus
* proximal left bronchial lesion
* anatomical abnormality of the bronchial tree
* suspicion of difficult mask ventilation or intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Rate of insertion | 300 seconds
  Rate of insertion, defined as successful placement of airway device in correct position without help of fibreoptic bronchoscopy

SECONDARY OUTCOMES:
Ease of use evaluated by the anesthesiologist | 3 hours
  Evaluation using a score (1 = easy to use, 2 = not so easy, 3 = difficult)
Quality of lung collapse | 3 hours
  Evaluation using a score (1 = atelectatic lung, 2 = lung well isolated but not atelectatic, 3 = failure of lung isolation)
Rate of misplacement occurring after patients removal from dorsal to lateral position | 1 hour
Rate of misplacement, occurring during surgery | 3 hours
Rate of requirement to a conventional double lumen tube | 3 hours
  ETView Double-Lumen Tube is not well positioned. It is withdrawn and replaced by a conventional double lumen tube

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Dumans-Nizard, MD, Principal Investigator — Hôpital Foch
Locations (1):
- Hopital Foch, Suresnes, France